CLINICAL TRIAL: NCT00284024
Title: Assessing the Feasibility of Testing Domperidone's Effect on Breastfeeding in Women With Insufficient Breast Milk: An RCT Pilot Study
Brief Title: Effectiveness of Domperidone to Increase Breastmilk Supply in Mothers With Low Supply
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: r05-60
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Insufficient Breastmilk Production
Keywords: breastfeeding; domperidone; efficacy; randomized controlled trial; compliance
MeSH Terms: conditions — Breast Feeding; Patient Compliance | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: domperidone

SUMMARY:
This study is testing if a medication called domperidone will help women produce more milk so that they can keep breastfeeding and not use formula. The study is also testing what dose of domperidone works best to increase breast milk production.

DETAILED DESCRIPTION:
Breastfeeding alone, until an infant is 6 months of age, is the best form of infant nutrition. There are many ways to help women breastfeed when they are having difficulties with the process, mostly involving support from a lactation consultant. However, some women, despite all appropriate non-medical interventions and support do not produce sufficient breast milk to meet the nutritional needs of their infant.

This is a feasibility study to determine how domperidone affects breast milk production in women with insufficient milk supply feeding term infants. This project will serve to refine and advance the design of a subsequent full-scale clinical trial.

The goal of this study is to: a) refine the intervention strategy (drug dosage), b) to define the target population and ensure adequate enrollment, c) assess protocol adherence and subject retention, and d) collect preliminary data to establish measures of clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

Women

* healthy women
* inadequate milk supply
* read/speak English

Infants

* healthy term infants (≥ 38 weeks gestational age)
* age ≥ 2wks and ≤3mths
* surpassed birth weight

Exclusion Criteria:

Mother

* cardiac anomalies
* breast or endocrine abnormalities (i.e. breast CA, pituitary adenomas)
* medications contraindicated with domperidone use
* drug or alcohol use
* use of hormonal contraception

Infant

* physical anomalies making breastfeeding difficult (i.e. cleft palate)
* cardiac anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
success of continuing breastfeeding
amount of supplementation used

SECONDARY OUTCOMES:
concentration of domperidone in milk
concentration of domperidone and prolactin in milk
maternal satisfaction
protocol adherence and barriers

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Ivanyi, MD, Principal Investigator — McMaster University
Locations (1):
- Stonechurch Family Health Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208